CLINICAL TRIAL: NCT00075803
Title: A Randomized Double-blind Trial of Fluconazole Versus Voriconazole for the Prevention of Invasive Fungal Infections in Allogeneic Blood and Marrow Transplant Patients (BMT CTN #0101)
Brief Title: Comparison of Fluconazole vs Voriconazole to Treat Fungal Infections for Blood and Marrow Transplants (BMT CTN 0101)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMTCTN0101; BMT CTN 0101 (Other: Blood and Marrow Transplant Clinical Trial Network); U01HL069294 (NIH); 5U24CA076518 (NIH); NCT00322088 (obsolete NCT alias)
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Results first posted 2015-09-04 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Lymphoma; Infection; Leukemia
Keywords: Myelodysplastic and Myeloproliferative Diseases
MeSH Terms: conditions — Lymphoma; Infections; Leukemia; Myelodysplastic-Myeloproliferative Diseases | interventions — Fluconazole; Voriconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluconazole (Active Comparator): The dose of fluconazole is 400 mg by mouth or intravenous drip.
  Interventions: Drug: Fluconazole
- Voriconazole (Experimental): The dose of oral voriconazole is 200 mg twice daily. When voriconazole must be given intravenously, it will be given at a dose of 200 mg every 12 hours for the duration of intravenous therapy.
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Fluconazole — Fluconazole will be administered orally once daily. Fluconazole capsules should be taken at least one hour before or one hour after a meal. If oral drug is not possible, it will be given intravenously once daily in a total volume of 200 mL in patients > 12 years. For adults, each 200 mL infusion will be administered over 2 hours. In patients < 12 years, intravenous doses will be prepared.
  Other Names: Diflucan
  Arms: Fluconazole
Drug: Voriconazole — Voriconazole will be administered orally twice daily. Voriconazole capsules should be taken at least one hour before or one hour after a meal. Taken concomitantly with food, bioavailability of voriconazole is reduced. If oral drug is not possible, it will be given intravenously at a dosage of 200 mg every 12 hours over two hours in patients > 12 years. Each voriconazole dose will be diluted to a total volume of 200 mL in patients > 12 years. Volumes of the formulation required to provide 4 mg/kg doses for children age < 12 years.
  Other Names: Vfend
  Arms: Voriconazole

SUMMARY:
The study is designed as a Phase III, randomized, double-blind, multicenter, prospective, comparative study of fluconazole versus voriconazole for the prevention of fungal infections in allogeneic transplant recipients. Recipients will be stratified by center and donor type (sibling vs. unrelated) and will be randomized to either the fluconazole or voriconazole arm in a 1:1 ratio.

DETAILED DESCRIPTION:
BACKGROUND:

Allogeneic blood and marrow transplant patients are highly susceptible to invasive fungal infection prior to engraftment, due to neutropenia and mucosal injury. After engraftment, an impairment of cell mediated immunity from graft-versus-host disease (GVHD) and the use of aggressive immunosuppressive therapies, such as corticosteroids, leave patients vulnerable to invasive fungal infections. Recipients of alternate donor transplants are especially susceptible due to slow reconstitution of cell mediated immunity.

Fluconazole prophylaxis in prospective randomized trials of both autologous and allogeneic transplant recipients has been demonstrated to reduce invasive fungal infections due to yeasts prior to engraftment. A prolonged course of fluconazole given during the first 75 days (to cover the early post-engraftment period of risk) is highly effective in the prevention of early and later yeast infections. This has translated into a survival benefit. A recent analysis of long-term outcomes of these individuals demonstrated a continuing benefit beyond the course of prophylaxis with a further benefit in survival. In another study of various factors associated with survival after matched unrelated donor transplants, fluconazole prophylaxis was an independent predictor for overall survival in a multivariate analysis. Fluconazole prophylaxis has been found to be effective and safe with few substantive drug interactions and has been widely adopted by transplant clinicians.

DESIGN NARRATIVE:

This is a randomized, double-blind, multicenter, prospective, comparative study of fluconazole versus voriconazole for the prevention of fungal infections in allogeneic hematopoietic transplant recipients and cord blood recipients in children under the age of 12. Prior to the start of the pre-transplant conditioning regimen, participants will give written informed consent and be screened for eligibility. Participants who meet all entry criteria will be assigned randomly to voriconazole or fluconazole within 72 hours of Day 0. Participants will begin the study drug on Day 0 (after completion of the conditioning regimen). Day 0 is defined as the day infusion of the stem cell product is completed. The study drug will be continued until Day 100 following transplant or until one or more criteria for early withdrawal are met. Continuation of the study drug beyond Day 100 is permitted for participants who meet specific criteria. The development of any fungal infection during prophylaxis will be classified according to the definitions listed in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Must receive an allogeneic peripheral blood or marrow transplant from a family or unrelated donor, or for children under the age of 12, a cord blood transplant from either a sibling or other donor
* Must have a 5 or 6 of 6 human leukocyte antigens (HLA)-matched donor. The match may be determined at serologic level for HLA-A and HLA-B loci. For sibling donors, matching may be determined at serologic level for HLA-DR; for unrelated donors, matching for HLA-DRB1 must be at the high-resolution molecular level
* Must have one of the following underlying diseases:

  1. Acute myelogenous leukemia (AML)
  2. Acute lymphocytic leukemia (ALL)
  3. Acute undifferentiated leukemia (AUL)
  4. Acute biphenotypic leukemia in first or second complete remission
  5. Chronic myelogenous leukemia (CML) in either chronic or accelerated phase
  6. One of the following myelodysplastic syndrome(s) (MDS):

     1. Refractory anemia
     2. Refractory anemia with ringed sideroblasts
     3. Refractory cytopenia with multilineage dysplasia
     4. Refractory cytopenia with multilineage dysplasia and ringed sideroblasts
     5. Refractory anemia with excess blasts-1 (5-10% blasts)
     6. Refractory anemia with excess blasts-2 (10-20% blasts)
     7. MDS, unclassified
     8. MDS associated with isolated del (5q)
     9. Chronic myelomonocytic leukemia (CMML)
  7. Lymphoma (including Hodgkin's) with chemosensitive disease (at least 50% response to chemotherapy) and receiving a related donor transplant
* Receiving myeloablative conditioning regimens
* Adequate physical function (cardiac, hepatic, renal, and pulmonary), within 6 weeks of initiation of conditioning (preferably within 4 weeks) unless otherwise specified
* Baseline galactomannan blood samples drawn within 30 days prior to randomization with the results available prior to randomization (72 hours prior to transplant)
* Chest computed tomography (CT) scans within 6 weeks prior to randomization if the results of the baseline galactomannan blood sample are not available prior to randomization (72 hours prior to transplant)

Exclusion Criteria:

* Invasive yeast infection within the 8 weeks prior to conditioning regimen initiation. Patients are eligible if colonized or have had superficial infection. Patients with a history of candidemia greater than 8 weeks prior to conditioning must have a negative blood culture within 14 days of conditioning (within 7 days is recommended), no clinical signs of candidemia, and may not still require antifungal therapy
* Presumptive, proven, or probable aspergillus or other mold infection or deep mycoses (including hepatosplenic candidiasis) within 4 months prior to conditioning regimen initiation
* Uncontrolled viral or bacterial infection at the time of study registration
* Pregnant or breastfeeding. Women of child-bearing age must avoid becoming pregnant while receiving antifungal agents
* Karnofsky performance status less than 70% or Lansky status less than 50% for patients under 16 years old unless approved by the medical monitor or protocol chair
* History of allergy or intolerance to azoles (e.g., fluconazole, itraconazole, voriconazole, posaconazole, ketoconazole, miconazole, clotrimazole)
* Requiring therapy with rifampin, rifabutin, carbamazepine, cisapride (Propulsid®), terfenadine (Seldane®), astemizole (Hismanal®), ergot alkaloids, long-acting barbiturates, or who have received more than 3 days treatment with rifampin or carbamazepine within 7 days prior to conditioning regimen initiation. Patients on therapeutic anticoagulation with coumadin (1 mg/day for port prophylaxis is permitted)
* Receiving sirolimus
* Prolonged QTc syndrome at study entry
* HIV positive
* Receiving another investigational drug unless cleared by the medical monitors
* Received a prior allogeneic or autologous transplant
* Active central nervous system disease
* On fungal prophylaxis during conditioning regimen (it is recommended that fungal prophylaxis be suspended once patient is enrolled)
* Prior cancer, other than resected basal cell carcinoma or treated carcinoma in-situ. Cancer treated with curative intent less than 5 years previously will not be allowed unless approved by the medical monitor or protocol chair. Cancer previously treated with curative intent over 5 years ago will be allowed

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2003-11; Primary Completion 2006-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (33):
- United States (33):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCSD Medical Center, La Jolla, California
  - Stanford Hospital and Clinics, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Johns Hopkins/SKCCC, Baltimore, Maryland
  - Dana Farber Cancer Institute/Brigham & Womens, Boston, Massachusetts
  - Dana Farber Cancer Institute/Children's Hospital of Boston, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute/BMT, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Kansas City Cancer Centers, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - Washington University/St. Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas/MD Anderson CRC, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Utah BMT/Univ of Utah Med School, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Wingard JR, Carter SL, Walsh TJ, Kurtzberg J, Small TN, Baden LR, Gersten ID, Mendizabal AM, Leather HL, Confer DL, Maziarz RT, Stadtmauer EA, Bolanos-Meade J, Brown J, Dipersio JF, Boeckh M, Marr KA; Blood and Marrow Transplant Clinical Trials Network. Randomized, double-blind trial of fluconazole versus voriconazole for prevention of invasive fungal infection after allogeneic hematopoietic cell transplantation. Blood. 2010 Dec 9;116(24):5111-8. doi: 10.1182/blood-2010-02-268151. Epub 2010 Sep 8. PMID 20826719
- [Result] Mauskopf J, Chirila C, Graham J, Gersten ID, Leather H, Maziarz RT, Baden LR, Bolanos-Meade J, Brown JM, Walsh TJ, Horowitz MH, Kurtzberg J, Marr KA, Wingard JR. Comparative cost-effectiveness analysis of voriconazole and fluconazole for prevention of invasive fungal infection in patients receiving allogeneic hematopoietic cell transplants. Am J Health Syst Pharm. 2013 Sep 1;70(17):1518-27. doi: 10.2146/ajhp120599. PMID 23943184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from November 2003 through September 2006
Groups:
- Fluconazole: fluconazole prophylaxis
- Voriconazole: voriconazole prophylaxis
Period: Overall Study
Arm/Group | Fluconazole | Voriconazole
Started | 295 | 305
Completed | 295 | 305
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluconazole | Voriconazole | Total
Number analyzed (Participants) | 295 | 305 | 600
Age, Customized [Median (Full Range); unit: years] | 43 [9 to 65] | 43 [3 to 66] | 43 [3 to 66]
Age, Customized [Number; unit: participants]
  <18 years | 24 | 27 | 51
  ≥18 years | 271 | 278 | 549
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 135 | 269
  Male | 161 | 170 | 331
Race/Ethnicity, Customized [Number; unit: participants]
  White | 265 | 276 | 541
  Other | 30 | 29 | 59
Graft Source [Number; unit: participants]
  Bone marrow | 109 | 106 | 215
  Peripheral blood | 186 | 197 | 383
  Cord blood | 0 | 2 | 2
Primary Disease [Number; unit: participants]
  Acute myeloid leukemia | 101 | 133 | 234
  Acute lymphoblastic leukemia | 64 | 58 | 122
  Chronic myelogenous leukemia | 60 | 43 | 103
  Myelodysplastic syndrome | 49 | 49 | 98
  Non-Hodgkin lymphoma | 21 | 22 | 43
Human Leukocyte Antigen (HLA) Match [Number; unit: participants] — Patients must have a 5 or 6 of 6 HLA-matched donor. The match may be determined at serologic level for HLA-A and HLA-B loci.
  participants
    6 of 6 | 282 | 293 | 575
    5 of 6 | 13 | 12 | 25
Karnofsky/Lansky Performance Status [Number; unit: participants] — Assesses patient self-perceived global quality of life and functioning (excellent, very good, good, fair, poor), where 100 equals perfect quality of life.
  participants
    90% - 100% | 249 | 268 | 517
    < 90% | 46 | 37 | 83

OUTCOME MEASURES:

1. Primary Outcome: Fungal-free Survival (Percentage of Participants Alive and Free From Proven, Probable, or Presumptive Invasive Fungal Infection) at 180 Days Post-transplant
Time Frame: 180 days
Population: All randomized patients were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Fluconazole | Voriconazole
Number analyzed (Participants) | 295 | 305
percentage of patients | 74.9 [69.6 to 79.5] | 78.2 [73.1 to 82.4]

2. Secondary Outcome: Frequency of Invasive Fungal Infections (IFI)
Description: Incidence of proven, probably, or presumptive IFI
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Fluconazole | Voriconazole
Number analyzed (Participants) | 295 | 305
percentage of patients | 13.7 [9.8 to 17.6] | 12.7 [9.0 to 16.4]

3. Secondary Outcome: Percentage of Patients With Invasive Fungal Infection at 100, 180, and 365 Days
Time Frame: 100, 180, and 365 days
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Fluconazole | Voriconazole
Number analyzed (Participants) | 295 | 305
percentage of patients
  100 days | 9.5 [6.2 to 12.8] | 5.6 [3.1 to 8.1]
  180 days | 11.2 [7.7 to 14.7] | 7.3 [4.4 to 10.2]
  365 days | 13.7 [9.8 to 17.6] | 12.7 [9.0 to 16.4]

4. Secondary Outcome: Overall Survival
Time Frame: 100, 180, and 365 days
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Fluconazole | Voriconazole
Number analyzed (Participants) | 295 | 305
percentage of patients
  100 days | 85.4 [80.9 to 89.0] | 90.1 [86.2 to 93.0]
  180 days | 80.0 [75.0 to 84.1] | 81.2 [76.3 to 85.1]
  365 days | 70.2 [64.6 to 75.1] | 67.8 [62.1 to 72.8]

5. Secondary Outcome: Relapse Free Survival
Time Frame: 100, 180, and 365 days
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Fluconazole | Voriconazole
Number analyzed (Participants) | 295 | 305
percentage of patients
  100 days | 83.1 [78.3 to 86.9] | 86.1 [81.7 to 89.6]
  180 days | 74.9 [69.6 to 79.5] | 73.9 [68.5 to 78.5]
  365 days | 63.3 [57.4 to 68.6] | 61.2 [55.5 to 66.5]

6. Secondary Outcome: Frequency of Use of Amphotericin B or Caspofungin
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Fluconazole | Voriconazole
Number analyzed (Participants) | 295 | 305
percentage of patients | 30.2 [24.9 to 35.5] | 24.1 [19.2 to 29.0]

7. Secondary Outcome: Duration of Use of Amphotericin B or Caspofungin
Time Frame: 180 days
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Fluconazole | Voriconazole
Number analyzed (Participants) | 295 | 305
days
  Number of days on study drug | 91 [27 to 100] | 96 [34 to 101]
  Start day of empiric antifungal therapy | 16 [10 to 33] | 12 [8 to 39]
  Days of empiric antifungal therapy | 7 [4 to 17] | 7 [5 to 15]

8. Secondary Outcome: Time to and Severity of Acute and Chronic Graft vs Host Disease (GVHD)
Time Frame: 100 and 365 days
Measure: Number; unit: participants
Arm/Group | Fluconazole | Voriconazole
Number analyzed (Participants) | 295 | 305
participants
  Acute GVHD grade II-IV at day 100 | 132 | 116
  Acute GVHD grade III-IV at day 100 | 42 | 27
  Chronic GVHD at 1 year | 138 | 137

9. Secondary Outcome: Utility of Galactomannan Assay in Diagnosis of Aspergillus and Response to Therapy
Description: Although there were 82 Galactomannan (GM) positives, 4 were excluded due to piperacillin/tazobactam administration, without other documentation of IFI, and were deemed false positives.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Fluconazole | Voriconazole
Number analyzed (Participants) | 295 | 305
participants
  GM+ | 43 | 35
  GM- | 252 | 270

10. Secondary Outcome: Time to Neutrophil Engraftment
Time Frame: 28 days
Reporting Status: Not Posted

11. Secondary Outcome: Time to Platelet Engraftment
Time Frame: 180 days
Reporting Status: Not Posted

12. Secondary Outcome: Failure to Engraft
Time Frame: day 42
Measure: Number; unit: participants
Arm/Group | Fluconazole | Voriconazole
Number analyzed (Participants) | 295 | 305
participants | 11 | 9

13. Secondary Outcome: Freedom From Possible, Presumptive, Probable, or Proven Invasive Fungal Infection, Death, or Withdrawal of Study Drug Due to Toxicity, Intolerance, or an Empirical Trial of Amphotericin B or Caspofungin Greater Than 14 Consecutive Days
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Fluconazole | Voriconazole
Number analyzed (Participants) | 295 | 305
participants
  IFI after relapse/progression | 2 | 8
  IFI before engraftment | 12 | 8
  IFI who had failure to engraft | 2 | 1
  IFI after aGVHD (grades II-IV) | 11 | 14
  IFI while on study drug (up to day 100) | 19 | 10
  IFI after premature withdrawal of study drug | 11 | 16
  IFI after start other prophylaxis (not study drug) | 8 | 11
  IFI after empiric therapy | 13 | 12

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Fluconazole | Voriconazole
Serious Adverse Events (participants affected / at risk) | 78/295 | 73/305
Other Adverse Events (participants affected / at risk) | 196/295 | 199/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluconazole (N=295) | Voriconazole (N=305)
Cardiovascular arrhythmia (Cardiac disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Pulmoary embolus (Vascular disorders) | 3 | 1
troponin level grade 4 (Congenital, familial and genetic disorders) | 1 | 0
hypotension (Vascular disorders) | 1 | 0
Guillian-Barre syndrome (Nervous system disorders) | 1 | 0
PTLD (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
acute renal failure (Renal and urinary disorders) | 1 | 0
confusion (Nervous system disorders) | 1 | 0
seizure (Nervous system disorders) | 1 | 0
hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
AV Block - third Degree (Cardiac disorders) | 0 | 1
Acute Mental Status Change (Psychiatric disorders) | 0 | 1
Urinary Frequency/urgency (Renal and urinary disorders) | 0 | 1
Elevated Magnesium (Investigations) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular Ischemia (Nervous system disorders) | 0 | 1
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 1
Sagittal Sinus Thrombosis (Nervous system disorders) | 0 | 1
Death at home, unexpected (General disorders) | 0 | 1
Pain, Site Right Kidney (Musculoskeletal and connective tissue disorders) | 0 | 1
Appendectomy (Surgical and medical procedures) | 0 | 1
Photopsia (Eye disorders) | 0 | 2
Somnolence (Nervous system disorders) | 6 | 5
Psychosis (Psychiatric disorders) | 2 | 1
Seizures (Nervous system disorders) | 0 | 1
Confusion (Nervous system disorders) | 4 | 5
EKG Abnormality (Cardiac disorders) | 8 | 5
Arrythmia (Cardiac disorders) | 10 | 7
Hypotension (Vascular disorders) | 16 | 16
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 3 | 2
Renal Failure (Renal and urinary disorders) | 10 | 7
Hemorrhagic Cystitis (Renal and urinary disorders) | 0 | 0
Hepatic Dysfunction (Hepatobiliary disorders) | 17 | 17
Mucositis/Stomatitis (Gastrointestinal disorders) | 11 | 16
Hemorrhage (Vascular disorders) | 12 | 9
HUS/TTP/thrombotic microangiopathy (Blood and lymphatic system disorders) | 6 | 4
Vascular Leak Syndrome (Vascular disorders) | 7 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 45 | 39
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 43 | 36
Allergic Reaction / Hypersensitivity (General disorders) | 0 | 0
Hypertension (Vascular disorders) | 0 | 0
Fever (General disorders) | 0 | 1
Rigors/Chills (General disorders) | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0
Vomitting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluconazole (N=295) | Voriconazole (N=305)
Photopsia (Eye disorders) | 18 | 19
Somnolence (Nervous system disorders) | 24 | 30
Psychosis (Psychiatric disorders) | 20 | 27
Seizures (Nervous system disorders) | 9 | 6
Confusion (Nervous system disorders) | 57 | 49
EKG Abnormality (Cardiac disorders) | 30 | 30
Arrhythmia (Cardiac disorders) | 4 | 7
Hypotension (Vascular disorders) | 24 | 9
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 8 | 1
Hemorrhagic Cystitis (Renal and urinary disorders) | 19 | 10
Hepatic Dysfunction (Hepatobiliary disorders) | 87 | 101
Liver Abnormality (Hepatobiliary disorders) | 17 | 12
Mucositis/Stomatitis (Gastrointestinal disorders) | 66 | 62
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 20 | 18
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 34 | 23
Allergic Reaction / Hypersensitivity (General disorders) | 5 | 5
Hypertension (Vascular disorders) | 7 | 4
Fever (General disorders) | 27 | 18
Rigors, chills (General disorders) | 14 | 3
Nausea (Gastrointestinal disorders) | 25 | 17
Vomiting (Gastrointestinal disorders) | 15 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2006-03-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT00075803/Prot_SAP_ICF_000.pdf